CLINICAL TRIAL: NCT04423471
Title: Neuroinflammation and Affective and Cognitive Symptoms in Patients Suffering From Major Depression and Psoriasis and Their Evolution With Treatment: A Prospective Study
Brief Title: Neuroinflammation, Affective and Cognitive Symptoms in Major Depression and Psoriasis
Acronym: INPSYDER
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PI-16-150
Record Dates: First submitted 2020-02-27; First posted 2020-06-09 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Psoriasis; Neuroinflammation; Major Depressive Disorder; Cognitive Symptom; Immunological Abnormality
Keywords: Neuroinflammation; Depression; Psoriasis
MeSH Terms: conditions — Psoriasis; Neuroinflammatory Diseases; Depressive Disorder, Major; Neurobehavioral Manifestations; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — A blood collection will be performed to collect serum and PBMC (peripheral blood mononuclear cells). Serum samples will be centrifuged at 1750 rpm for 10 minutes, the supernatant will be collected and frozen at -20 ° C. For PBMC, Ficoll gradient centrifugation of blood samples with anticoagulant will be carried out. Once the PBMCs are separated, they will be frozen with 20% DMSO in RPMI culture doctor with 20% fetal calf serum (FCS) and stored in liquid nitrogen. Blood samples will also be obtained for the total extraction of RNA with 3 ml of Paxgene® tubes, processed and frozen at -80 ° C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Psoriasis patients who will receive systemic treatment (mainly methotrexate)
  Interventions: Diagnostic Test: Sociodemographic variables
- Group 2: Psoriasis patients who will receive a biological treatment
  Interventions: Diagnostic Test: Sociodemographic variables
- Group 3: Patients with major depression who will receive an antidepressant treatment
  Interventions: Diagnostic Test: Sociodemographic variables

INTERVENTIONS:
Diagnostic Test: Sociodemographic variables — * Sociodemographic variables: Sex / Age / Marital status / Level of studies completed / Employment status.
  * General clinical variables: Body mass index (BMI), Medical comorbidities and Charlson Comorbidity Index, Active drug treatments
  * Clinical psoriasis variables: BSA, PASI, ScalpPASI, PPPASI, DLQI, time since the diagnosis of psoriasis, previous treatments for psoriasis.
  * Clinical depression variables: Psychiatric diagnoses according to clinical interview and DSM-5 criteria, age of onset and time of evolution from the first episode of major depression, time of evolution of the current episode of major depression, previous treatments for depression.
  * Psychopathological variables: HADS, PHQ-9, MADRS, GAD-7, SHAPS, The Irritability Questionnaire, PSS, FSS, MoCA.
  * Immunological and biochemical variables: Acute phase biomarkers, Proinflammatory cytokines, Anti-inflammatory cytokines, HPA axis, Microglia activation, Neurogenesis.
  * Result variables: Changes in PASI or MADRS scores
  Other Names: General clinical variables; Clinical psoriasis variables; Clinical depression variables; Psychopathological variables; Immunological and biochemical variables; Result variables

SUMMARY:
Objectives: To identify peripheral neuroinflammatory markers in patients suffering from major depression or psoriasis in relation to affective symptoms (anxiety, depression, irritability), fatigue and cognitive symptoms; and their change after specific treatments.

Methodology: Observational prospective cohort study in patients diagnosed with major depression and patients with plaque psoriasis, who naturalistically undergo different treatments (systemic or biological for psoriasis, antidepressants for depression). Forty-one patients with major depression attending psychiatric consultations and 82 patients with psoriasis attending dermatology consultations at Hospital Universitari Germans Trias i Pujol aged 18 to 65 years old will be selected for inclusion. All of them will be assessed at baseline and after 4 months treatment through a series of demographic and clinical variables, psychiatric diagnosis, psychopathological scales and immunological and biochemical variables after blood draw for obtaining serum, peripheral blood mononuclear cell (PBMC) and extraction of total RNA. Investigators will analyze the correlation between immunological markers and affective and cognitive symptoms at baseline, as well as their variation after treatment. Subsequently, a bivariate comparative analysis will be carried out, where statistically significant or marginally significant variables associated with psychopathological variables will be used to construct a multivariate model of binary logistic regression.

DETAILED DESCRIPTION:
Design This is a prospective observational study of cohorts with patients diagnosed with major depression or psoriasis and subjected to different treatments with systemic or biological drugs in the case of psoriasis, and with antidepressants in the case of major depression.

Subjects of study The subjects that will participate in this study will be outpatients treated in the Dermatology Consultations and the Psychiatric Consultations of the Germans Trias i Pujol University Hospital (Badalona, Spain), clinically diagnosed with psoriasis or major depression.

Inclusion criteria:

* Age between 18 and 65
* Clinical diagnosis of 1) In the psoriasis group: diagnosis of plaque psoriasis made by a dermatologist, lasting at least 6 months; 2) In the major depression group: clinical diagnosis of major depression according to DSM-5 criteria made by a psychiatrist.
* Patients receiving systemic or biological treatment for psoriasis, or antidepressant for major depression.

Exclusion criteria:

* Previous treatments for psoriasis: narrow band ultraviolet B radiation (NBUBR) phototherapy in the last 2 weeks; Psoralene+ultraviolet A (PUVA) phototherapy in the last 4 weeks; conventional systemic treatments in the last 4 weeks; biological treatments in the last 3 months
* Previous antidepressant treatments in the last 6 weeks
* Antipsychotic or eutimizing treatments in the last 6 weeks
* The presence of concurrent psychotic symptoms
* Alcohol or drug use disorders, with active consumption during the last 3 months
* Pregnant women
* Serious and / or unstable medical disorders, Addison or Cushing's disease, Rheumatoid arthritis or systemic lupus erythematosus.

Patients will be assigned to three groups:

* Group 1 - psoriasis patients who will receive systemic treatment (mainly methotrexate)
* Group 2 - psoriasis patients who will receive a biological treatment
* Group 3 - patients with major depression who will receive an antidepressant treatment

Sample's size calculation The required sample size has been calculated based on the possible differences in the biomarkers: C reactive protein (CRP), interleukin IL-6, etc. Accepting an alpha risk of 0.05 and a beta risk of less than 0.2 in a bilateral contrast, 41 subjects are needed in each of the three groups to detect a difference equal to or greater than 2/3 of the standard deviation. A follow-up loss rate of 10% has been estimated. Therefore, a total of 123 patients will be evaluated.

Variables

* Sociodemographic variables: Sex / Age / Marital status / Level of studies completed / Employment status
* General clinical variables

  * Body mass index (BMI)
  * Medical comorbidities and Charlson Comorbidity Index
  * Active drug treatments
* Clinical psoriasis variables

  * BSA (Body Surface Area). Calculation of the body surface covered by injuries.
  * PASI (Psoriasis Area and Severity Index). It is a measure of the severity and overall coverage of psoriasis. All calculations are combined in a single score in the range of 0 (absence of lesions) to 72 (the most severe case of psoriasis). Similarly, ScalpPASI (PASI applied to the scalp) and PPPASI (PASI applied to palmoplantar regions) will be calculated.
  * DLQI (Dermatology Life Quality Index). This instrument consists of 10 questions covering six domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships and concern for the treatment of psoriasis)
  * Time since the diagnosis of psoriasis
  * Previous treatments for psoriasis
* Clinical depression variables

  * Psychiatric diagnoses according to clinical interview and Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria (Structured Clinical Interview for DSM-5 (SCID-5).
  * Age of onset and time of evolution from the first episode of major depression
  * Time of evolution of the current episode of major depression
  * Previous treatments for depression
* Psychopathological variables

  * HADS (Hospital Anxiety and Depression Scale)
  * PHQ-9 (Patient Health Questionnaire)
  * MADRS (Montgomery Asberg Depression Rating Scale)
  * GAD-7 (Generalized Anxiety Disorder 7-item scale)
  * SHAPS (Snaith-Hamilton Pleasure Scale)
  * The Irritability Questionnaire
  * PSS (Perceived Stress Scale)
  * FSS (Fatigue Severity Scale)
  * MoCA (The Montreal Cognitive Assessment)
* Immunological and biochemical variables:

  * Acute phase biomarkers: C Reactive Protein (CRP)
  * Proinflammatory cytokines: IL-1β, IL-6, TNF-α, IL-12, IL-23, IL-17
  * Anti-inflammatory cytokines: IL-10, IL-4, Transforming growth factor-β (TGF-β)
  * Hypothalamus-pituitary-adrenal axis (HPA): Cortisol
  * Oxidative and nitrosative stress: Zinc, Glutathione, Albumin, Uric acid, Bilirubin
  * Microglia activation: miR-155, miR-126, miR223, miR146a, miR-21, miR-124
  * Neurogenesis: Brain-derived neurotrophic factor (BDNF) in serum
  * Lymphocyte subpopulations in peripheral blood (Th1, Th2, Th17, Th1 / 17, Treg, ship cells, central memory and effector memory)
* Result variables:

  * Response to treatment (changes in PASI or MADRS scores)

Data collection and analysis All outpatients with the diagnosis of psoriasis attended in the Dermatology Consultations of the Germans Trias i Pujol Hospital, as well as all those patients with the diagnosis of major depression treated in the Psychiatric Consultations of the same center, will be evaluated for the recruitment.

* Recruitment visit: It will be performed by one of the dermatologists (in the psoriasis group) or by one of the psychiatrists (in the major depression group) participating in the study. The patient will be informed about the study and their written consent will be requested. Subsequently, the inclusion and exclusion criteria will be reviewed, and all demographic and clinical variables will be collected.
* Baseline visit: A blood collection will be performed to collect serum and PBMC (peripheral blood mononuclear cells). Serum samples will be centrifuged at 1750 rpm for 10 minutes, the supernatant will be collected and frozen at -20 ° C in the Immunology Laboratory of the Germans Trias i Pujol Institute. For PBMC, Ficoll gradient centrifugation of blood samples with anticoagulant will be carried out. Once the PBMCs are separated, they will be frozen with 20% dimethyl sulfoxide (DMSO) in Roswell Park Memorial Institute (RPMI) culture doctor with 20% fetal calf serum (FCS) and stored in liquid nitrogen in the Cryobiology Platform of the Germans Trias i Pujol Institute. Blood samples will also be obtained for the total extraction of RNA with 3 ml of Paxgene® tubes, processed and frozen at -80 ° C in the immunology laboratory / Also in this baseline visit, one of the psychiatrists will visit the patient and apply the interview semi-structured clinic and psychopathological evaluation questionnaires.
* Follow-up visit after 16 weeks of treatment: Clinical variables will be collected and the same procedures as during the baseline visit will be performed.

Statistical analysis First, a descriptive analysis of the sample will be carried out. Categorical variables will be summarized with frequencies and percentages, while quantitative variables will be described with the mean and standard deviation if they have a normal distribution, or the median and the 25th and 75th percentiles otherwise.

Secondly, the correlation between the severity of psoriasis (PASI) at the baseline visit (in all patients) and the different scores of the psychopathological scales will be analyzed. Since the PASI does not follow a normal distribution, it will be carried out with the Spearman linear correlation test (Spearman rho).

Subsequently, a bivariate comparative analysis between the analytical and psychopathological variables will be carried out. Categorical variables will be compared with Fisher's square or exact Chi test, according to the application conditions, and quantitative variables with the Student's T test for independent data or the non-parametric Mann-Whitney U test. The statistically significant or marginally significant variables (P <0.01) associated with psychopathological variables in the bivariate analysis will be used to construct a multivariate model of binary logistic regression, in order to evaluate the joint factors with greater discrimination capacity of each of the psychopathological variables. For the model, the odds ratio will be displayed along with its 95% confidence intervals and the model calibration will be evaluated with the Hosmer and Lemeshow test and its ability to discriminate using Receiver Operating Characteristic (ROC) curves. In all cases, P values below 0.05 will be considered statistically significant. The analysis will be carried out with the SPSS 22.0 software.

Limitations of the study The study is conducted in a tertiary referral hospital, so the sample of patients with psoriasis or major depression may not be representative of the general population of patients with these diseases.

Psychopathological measures are carried out through fully validated questionnaires in Spanish in different population samples, including populations with comorbid medical conditions, but not specifically in patients with psoriasis, except for DLQI.

Patients with psoriatic arthritis, although with high levels of inflammation, are likely to be on chronic treatment with anti-inflammatory drugs that may affect the results. In any case, the use of these treatments will be used as a covariate.

Ethical aspects The project will be submitted to the Ethical Research Committee (ERC)-Germans Trias i Pujol University Hospital for approval. Subjects will be included once they have given their informed consent. The ethical principles of the Declaration of Helsinki (Fortaleza, 2013), the Standards of Good Clinical Practice, the legislation on biomedical research (Law 14/2007), the obtaining and processing of biological samples and biobanks (RD 1716) will be respected. / 2011) and clinical trials with medications (RD 1090/2015). The data will be processed in accordance with Organic Law 15/1999, on the Protection of Personal Data.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Clinical diagnosis of:

  * In the psoriasis group: diagnosis of plaque psoriasis made by a dermatologist, lasting at least 6 months.
  * In the major depression group: clinical diagnosis of major depression according to DSM-5 criteria made by a psychiatrist.
* Patients receiving systemic or biological treatment for psoriasis, or antidepressant for major depression.

Exclusion criteria:

* Previous treatments for psoriasis

  * UVBBE phototherapy in the last 2 weeks
  * PUVA phototherapy in the last 4 weeks
  * Conventional systemic treatments in the last 4 weeks
  * Biological treatments in the last 3 months
* Previous antidepressant treatments in the last 6 weeks
* Antipsychotic or eutimizing treatments in the last 6 weeks
* The presence of concurrent psychotic symptoms
* Alcohol or drug use disorders, with active consumption during the last 3 months
* Pregnant women
* Serious and / or unstable medical disorders, Addison or Cushing's disease, Rheumatoid arthritis or systemic lupus erythematosus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects that will participate in this study will be outpatients treated in the External Dermatology Consultations and the External Psychiatric Consultations of the Germans Trias i Pujol University Hospital (Badalona, Spain), clinically diagnosed with psoriasis or major depression.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between immunological markers and affective and cognitive symptoms at baseline. | Baseline
  To evaluate the relationship of psychiatric symptoms (affective symptoms, fatigue, cognitive deficits) and markers of inflammation, HPA axis, oxidative and nitrosative stress, gliosis and neurogenesis in both groups of psoriasic and depressive patients.
Changes in immunological markers and affective and cognitive symptoms between baseline and after 4 months of treatment. | Baseline and at 4 months
  To evaluate the changes of psychiatric symptoms (affective symptoms, fatigue, cognitive deficits) and markers of inflammation, HPA axis, oxidative and nitrosative stress, gliosis and neurogenesis, after treatment for psoriasis with systemic or biological treatment of psoriasis and with antidepressant treatment for major depression.

SECONDARY OUTCOMES:
Correlation between immunological markers and the course of psychiatric comorbidity in relation to anti-inflammatory treatments | Baseline and at 4 months
  To assess the relationship between the variations of the biological markers of inflammation, HPA axis, oxidative and nitrosative stress, gliosis and neurogenesis and the course of psychiatric comorbidity in relation to the different anti-inflammatory treatments for psoriasis.
Correlation between the course of major depression with antidepressant treatment and biomarkers of inflammation | Baseline and at 4 months
  To evaluate the relationship between the course of major depressive illness with treatment and biomarkers of inflammation, HPA axis, oxidative and nitrosative stress, gliosis and neurogenesis

CONTACTS AND LOCATIONS:
Overall Officials: Crisanto Díez-Quevedo, MD, PhD, Study Chair — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia, Spain